CLINICAL TRIAL: NCT01631721
Title: Affective Influences on Adolescent Sexual Risk Behavior: Couple & Family Contexts
Brief Title: Couple & Family Contexts
Acronym: CFC
Status: Completed | Type: Observational
Sponsor: New York University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: NICHD_064734; R01HD064734 (NIH)
Record Dates: First submitted 2012-06-26; First posted 2012-06-29 (Estimated); Last update posted 2022-10-28 (Actual); Status verified 2016-03

CONDITIONS: Behavior and Behavior Mechanisms
Keywords: adolescent couple decision-making; parenting practices; sexual risk behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Cohort 1: Cohort of adolescents recruited in 2012-2013 of study
- Cohort 2: Cohort of adolescents recruited in year 2013-2014 of study
- Cohort 3: Cohort of adolescents recruited in year 2014-15 of study

SUMMARY:
The purpose of this study is to understand the factors that lead to adolescent sexual risk behavior by investigating both the family contexts and romantic relationships that influence adolescent couples' decision-making.

DETAILED DESCRIPTION:
In the United States, inner-city African American and Latino youth are vulnerable to the negative consequences of sexual risk behavior. Despite the fact that sexual risk behavior is a dyadic behavior, almost all of the social-cognitive theories emphasize individual-based variables to explain behavior. Little research has studied both members of an adolescent couple or has used measures from each member to predict future sexual activity of that dyad. The overall aim of the present study is to identify explanatory models of couple sexual risk behavior among a sample of unmarried, non co-habiting Latino and African American high school-aged dyads that are romantically linked. In addition, the present research also will study the parents of adolescent couples. In doing so, the present research will apply theories of cognition, emotion and emotion regulation, and a new theory of parental monitoring to the study of adolescent sexual risk behavior among couples.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents must be between the ages of 17-19
* Adolescents must currently reside in the Bronx, New York
* Adolescents must be of Latino or African American descent
* Adolescents must identify as being currently involved in romantic relationship
* Adolescent and parent must both agree to being a participant
* Adolescent and parent must be able to participate in questionnaire activities

Exclusion Criteria:

* Any cognitive or psychiatric disability that would prevent successful participation of adolescent or parent in questionnaire activities

Ages: 17 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Latino and African American adolescents currently involved in romantic relationships who reside in the Bronx, New York.
Sampling Method: Probability Sample
Enrollment: 2960 (Actual)
Dates: Start 2010-11; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Incidence of vaginal intercourse with romantic partner | Baseline
  Number of times ever had vaginal intercourse with current romantic partner

SECONDARY OUTCOMES:
Frequency of condom use during vaginal intercourse with romantic partner | Baseline
  Of the number of times participant has ever had vaginal sex with romantic partner, number of times used a condom
Incidence of oral sex with romantic partner | Baseline
  Number of times has ever given/received oral sex with current romantic partner
Frequency of condom use for oral sex with romantic partner | Baseline
  Of number of times has ever had oral sex with current romantic partner, number of times used a condom
Incidence of anal intercourse with current romantic partner | Baseline
  Number of times has ever had anal intercourse with current romantic partner
Frequency of condom use for anal intercourse with romantic partner | Baseline
  Of times has ever had anal intercourse with current romantic partner, number of times used a condom
Frequency of condom use during vaginal intercourse with romantic partner | 6 Months Follow-up
  Of the number of times participant has ever had vaginal sex with romantic partner, number of times used a condom
Incidence of oral sex with romantic partner | 6 Months Follow-up
  Number of times has ever given/received oral sex with current romantic partner
Frequency of condom use for oral sex with romantic partner | 6 Months Follow-up
  Of number of times has ever had oral sex with current romantic partner, number of times used a condom
Incidence of anal intercourse with current romantic partner | 6 Months Follow-up
  Number of times has ever had anal intercourse with current romantic partner
Frequency of condom use for anal intercourse with romantic partner | 6 Months Follow-up
  Of times has ever had anal intercourse with current romantic partner, number of times used a condom
Incidence of vaginal intercourse romantic partner | 6 Months Follow-up
  Number of times ever had vaginal intercourse with current romantic partner

CONTACTS AND LOCATIONS:
Locations (1):
- Silver School of Social Work, New York University, New York, New York, United States